CLINICAL TRIAL: NCT06264258
Title: Evaluating Game-based Pediatric Diabetes Education
Brief Title: Game-based Pediatric Diabetes Education
Acronym: DVx-T1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rema Padman, Trustees Professor of Management Science & Healthcare Informatics, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY2023_00000285
Record Dates: First submitted 2024-02-12; First posted 2024-02-16 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1; Behavior, Health
Keywords: app; game; children; pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Health Behavior; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The investigators propose to conduct a longitudinal randomized controlled trial (RCT) over a 3-month period with a study population of 80 participants (40 in each arm) of 6-12 years old youth with type 1 diabetes (T1D).The investigators will quantify the impact of the mobile game app vs. standard care on T1D control (assessed by glycosylated hemoglobin or HbA1c measured during clinic visits and continuous glucose monitoring (CGM) parameters), physical activity levels and food choices of children (measured using food logs and surveys).
  The study will also assess changes in children's knowledge about the measured outcomes and investigate the feasibility and acceptability of game adoption and the barriers and challenges faced by patients, families and clinicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DVx-T1D+Standard Care (Experimental): Participants will continue receiving the clinic's standard of care. Anthropometrics, clinical and laboratory data will be collected at three time points, baseline, 6 weeks and 3 months. Participants will be asked to maintain food, glucose, and activity logs. In addition, participants in this arm will be provided a tablet that has the gaming applications already loaded and receive training on the application. Exposure time will be tracked by the application.
  Interventions: Behavioral: DVx-T1D™ app
- Standard Care (No Intervention): Participants will receive the clinic's standard of care. Anthropometrics, clinical and laboratory data will be collected at three time points, baseline, 6 weeks and 3 months. Participants will be asked to maintain food, glucose, and activity logs.

INTERVENTIONS:
Behavioral: DVx-T1D™ app — The intervention group will be introduced to the DVx-T1D™ app and the participants will go home with the tablets that has the game installed. Participants will be asked to play the game for 20 mins or more daily. The aim of the app is to impart good behavioral changes in children with T1D in terms of diabetes education, on how to treat a low or a high blood sugar event and make healthy eating choices.
  Arms: DVx-T1D+Standard Care

SUMMARY:
The goal of this study is to evaluate the impact of a mobile app video game called Digital Vaccine for Type 1 Diabetes (DVx-T1D)™, proposed as a low-risk, non-invasive, digital therapeutic candidate for behavior change in children 6 to 12 years of age with Type 1 Diabetes (T1D).

The investigators hypothesize that adoption of DVx-T1D™ by T1D patients will positively influence healthy dietary and physical activity behaviors by providing nutrition and lifestyle education through a playful, Artificial Intelligence (AI)-based, cartoon-style medium of mobile gaming, and result in improvements in their T1D control. The investigators propose to conduct a longitudinal randomized controlled trial (RCT) over a 3-month period with a study population of 80 T1D participants (40 each in two arms of the trial) of 6-12 years old. The investigators will quantify the impact of the mobile game app plus standard care vs. standard care (with no exposure to the app) on T1D control (assessed by glycosylated hemoglobin or HbA1c measured during clinic visits and continuous glucose monitoring (CGM) parameters measured at home), physical activity levels and food choices of children (measured using food logs and surveys). Game telemetry, food logs, clinical, anthropometric, demographic, and survey data will be collected to obtain adequately powered, theory-driven evidence of the value of game-based approaches delivered via mobile apps.

DETAILED DESCRIPTION:
Youth with T1D who comply with inclusion criteria and provide consent will be randomized to either the treatment arm (will be given a tablet with the game) or the control arm (no tablet will be given, no exposure to the game). Participants in both arms will continue receiving standard of care treatment. Participants will be asked to maintain food and activity logs and answer questionnaires about lifestyle.

Participants will be evaluated at baseline and at 3 months with interim contact in between. Devices will be downloaded to collect app usage data (game telemetry). Exposure time will be tracked by the application. Survey to elicit barriers and challenges encountered during the study will also be conducted.

ELIGIBILITY:
For youth:

* Be between the age of 6 to 12 years.
* Have been diagnosed with type 1 diabetes for at least 1 year.
* Be currently taking insulin through multiple daily injections or an insulin pump.
* Check blood sugar with a meter at least 4 times per day or use a continuous glucose monitor.
* Be willing to comply with all study visits and procedures.

For Parent:

* Biological or adopted parent with custody and medical decision making of the patients
* Living with identified patients
* Over 18 years old
* Resident of Allegheny County

Exclusion Criteria:

-Children with type 2 diabetes, cystic fibrosis related diabetes, or secondary diabetes.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c values and and insulin dose adjusted HbA1c before and after the intervention | Three months
  Change in HbA1C level and insulin dose adjusted HbA1c from baseline to 3 months.
Change in glucose average and variability | Three months
  Change in glucose average and variability as assessed by mean glucose and standard deviation (SD) as well as other continuous glucose monitor (CGM) parameters for those using this device.

SECONDARY OUTCOMES:
Changes in the quality of food consumption | Three months
  Changes in the quality of food consumption by comparing patients' food logs before and after the intervention, reported food choices and physical activity levels in the logs and surveys, and T1D specific diet and physical activity knowledge (for both participants and their parents).
Change in game play patterns over time | Three months
  Game play patterns learned from telemetry data over the 3 months of the experiment will be tracked and used to relate to the outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States